CLINICAL TRIAL: NCT03918239
Title: A Randomized, Open-label, Single-dose, Parallel-arm, Single-center, Phase 1 Study to Determine the Bioavailability of Lanadelumab Administered Subcutaneously With the Prefilled Syringe and the Autoinjector in Healthy Adult Volunteer Subjects
Brief Title: A Study to Determine the Bioavailability of Lanadelumab (SHP643) Administered Subcutaneously With the Prefilled Syringe and the Autoinjector in Healthy Adult Volunteer Participants.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHP643-102
Record Dates: First submitted 2019-04-15; First posted 2019-04-17 (Actual); Results first posted 2020-12-08 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-11

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — lanadelumab; rhoA GTP-Binding Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SHP643 Prefilled Syringe (PFS) (Experimental): Participants will receive 300 milligram (mg) of SHP643 PFS Subcutaneous (SC) injection into the abdomen on Day 1 during the in-house period (Day 1 to Day 5).
  Interventions: Drug: SHP643
- SHP643 Autoinjector (AI) (Experimental): Participants will receive 300 mg of SHP643 AI SC injection into the abdomen on Day 1 during the in-house period (Day 1 to Day 5).
  Interventions: Drug: SHP643

INTERVENTIONS:
Drug: SHP643 — Participants will receive injection of SHP643.
  Other Names: DX-2930 (formerly); Lanadelumab

SUMMARY:
The purpose of this study is to evaluate bioavailability of lanadelumab (SHP643) following a single, 2 milliliter (mL) subcutaneous (SC) dose of 300 milligrams (mg) delivered by prefilled syringe (PFS) or auto injector (AI) in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* An understanding, ability, and willingness to fully comply with study procedures and restrictions.
* Ability to voluntarily provide written, signed, and dated informed consent to participate in the study.
* Age 18-55, inclusive, at the time of consent. The date of signature of the informed consent is defined as the beginning of the screening period. This inclusion criterion will only be assessed at the first screening visit.
* Male, or non-pregnant, non-lactating female who agrees to comply with any applicable contraceptive requirements of the protocol or females of non-childbearing potential.
* Must be considered "healthy", per the investigator. Healthy status is defined by absence of evidence of any active or chronic disease following a detailed medical and surgical history, a complete physical examination including vital signs, 12-lead electrocardiogram (ECG), hematology, blood chemistry, and urinalysis.
* Body mass index between 18.5-33 kilogram per square meter (kg/m^2), inclusive, with a body weight greater than or equal to (>=) 45 kilogram (kg) (99 pounds [lbs]). This inclusion criterion will only be assessed at the screening visit and on Day -1.
* Willing and able to consume standardized meals during the confinement period of the study.
* All participants will be required to consume the identical meals on study days when serial PK blood samples are collected

Exclusion Criteria:

* Per the investigator, a history of any hematological, hepatic, respiratory, cardiovascular, renal, neurological or psychiatric disease, gall bladder removal, or current or recurrent disease that could affect the action, absorption, or disposition of the investigational product, or clinical or laboratory assessments.
* Per the investigator, a current or relevant history of physical or psychiatric illness, any medical disorder that may require treatment or make the participant unlikely to complete the study, or any condition that present's undue risk from the investigational product or procedures.
* Known or suspected intolerance or hypersensitivity to the investigational product, closelyrelated compounds, or any of the stated ingredients.
* Significant illness, as judged by the investigator, within 2 weeks of the dose of investigational product.
* Known history of alcohol or other substance abuse within the last year, per the investigator.
* Donation of blood or blood products (e.g. plasma or platelets) within 60 days prior to receiving the dose of investigational product.
* Within 30 days prior to the dose of investigational product.

  1. Have used an investigational product (if elimination half-life is <6 days, otherwise 5 half lives).
  2. Have been enrolled in a clinical study (including vaccine studies) that, in the investigator's opinion, may impact this Shire-sponsored study.
* Confirmed systolic blood pressure (BP) >139 millimeters of mercury (mmHg) or <89 mmHg, and diastolic BP >89 mmHg or <49 mmHg.
* Twelve-lead ECG values demonstrating QTcF >450 milliseconds (msec) (males) or >470 msec (females) at the screening visit or Day -1. If QTcF exceeds 450 msec (males) or 470 msec (females), the ECG should be repeated 2 more times and the average of the 3 QTcF values should be used to determine the participants eligibility.
* Positive screen for drugs of abuse and/or disallowed drugs (i.e. amphetamines, benzodiazepines, barbiturates, cocaine, opiates, phencyclidine) at screening, or drugs of abuse or alcohol on Day -1. This screen will include marijuana.
* Male participants who consume more than 21 units of alcohol per week or 3 units per day. Female participants who consume more than 14 units of alcohol per week or 2 units per day. One alcohol unit=1 beer or 1 wine (5 ounces [oz) per 150 milliliter [mL]) or 1 liquor (1.5 oz/40 mL) or 0.75 oz alcohol.
* Positive human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) antibody screen.
* Use of tobacco in any form (e.g. smoking or chewing) or other nicotine-containing products in any form (e.g. gum, patch, electronic). Ex-users must report that they have stopped using tobacco for at least 30 days prior to receiving the dose of investigational product.
* Routine consumption of more than 2 units of caffeine per day or participants who experience caffeine withdrawal headaches. One caffeine unit is contained in the following items: one 6 oz (180 ml) cup of coffee, two 12 oz (360 ml) cans of cola, one 12 oz cup of tea, and three 1 oz (85 g) chocolate bars. Decaffeinated coffee, tea, or cola are not considered to contain caffeine).
* Current use of any medication (including over-the-counter, herbal, or homeopathic preparations; with the exception of stable hormonal replacement therapy or hormonal contraceptives). Current use is defined as use within 14 days of the dose of investigational product. (Prior and Concomitant Treatment) for a list of permitted medications.
* Abnormal laboratory values considered clinically significant, as determined by the investigator, at screening or Day -1.
* History of any clinically significant surgery or procedure within 8 weeks of receiving the dose of investigational product, as determined by the investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 190 (Actual)
Dates: Start 2019-05-14 (Actual); Primary Completion 2019-11-13 (Actual); Study Completion 2019-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (1):
- Clinical Pharmacology of Miami, LLC, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fdc4db2bf003ab472e3

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at a single site in United States of America from 14 May 2019 (first participant first visit) to 13 November 2019 (last participant last visit).
Pre-assignment Details: A total of 190 participants were enrolled and received the treatment. Out of which, 173 participants completed this study.
Groups:
- SHP643 Prefilled Syringe (PFS): Participants received 300 milligram (mg) of SHP643 PFS Subcutaneous (SC) injection into the abdomen on Day 1 during the in-house treatment period (Day 1 to Day 5).
- SHP643 Autoinjector (AI): Participants received 300 mg of SHP643 AI SC injection into the abdomen on Day 1 during the in-house treatment period (Day 1 to Day 5).
Period: Overall Study
Arm/Group | SHP643 Prefilled Syringe (PFS) | SHP643 Autoinjector (AI)
Started | 94 | 96
Completed | 84 | 89
Not Completed | 10 | 7
Not completed — Lost to Follow-up | 3 | 1
Not completed — Pregnancy | 0 | 2
Not completed — Withdrawal by Subject | 3 | 3
Not completed — positive urine drug screening results | 4 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set consisted of all randomized participants who received the dose of SHP643.
Groups:
- Total: Total of all reporting groups
Arm/Group | SHP643 Prefilled Syringe (PFS) | SHP643 Autoinjector (AI) | Total
Number analyzed (Participants) | 94 | 96 | 190
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.6 (10.04) | 42.1 (9.67) | 40.8 (9.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 55 | 96
  Male | 53 | 41 | 94
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 91 | 92 | 183
  Not Hispanic or Latino | 3 | 4 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 19 | 32
  White | 81 | 77 | 158
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration Versus Time Curve From Time Zero to the Last Quantifiable Concentration (AUC0-last) of SHP643 in Plasma
Description: AUC(0-last) of SHP643 in plasma was reported. Geometric mean and geometric coefficient of variation percent (CV%) was reported.
Time Frame: Pre-dose, 8, 24, 48, 72, 96, 168, 336, 504, 672, 1008, 1344, 2016, 2664 hours post dose
Population: Pharmacokinetic (PK) set was defined as all randomized participants who received the complete dose of SHP643 and had sufficient data to calculate at least one primary PK endpoint. Here, the number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*microgram per milliliter (day*ug/mL)
Arm/Group | SHP643 Prefilled Syringe (PFS) | SHP643 Autoinjector (AI)
Number analyzed (Participants) | 89 | 89
day*microgram per milliliter (day*ug/mL) | 348.9 (33.4) | 376.5 (41.3)
Statistical Analysis 1: Comparison: SHP643 Prefilled Syringe (PFS) vs SHP643 Autoinjector (AI); An analysis of variance was performed with the natural log-transformed PK parameters as the dependent variable and treatment group as a fixed effect variable; Test type: Other — Analysis was performed for estimation of least square means only. Descriptive statistical analysis was the main analysis; ANOVA; Ratio of Geometric least squares Means = 1.079, 90% CI 2-sided [0.986 to 1.181]

2. Primary Outcome: Area Under the Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUC0-Inf) of SHP643 in Plasma
Description: AUC(0-infinity) of SHP643 in plasma was reported. Geometric mean and geometric coefficient of variation percent (CV%) was reported.
Time Frame: Pre-dose, 8, 24, 48, 72, 96, 168, 336, 504, 672, 1008, 1344, 2016, 2664 hours post-dose
Population: PK set was defined as all randomized participants who received the complete dose of SHP643 and had sufficient data to calculate at least one primary PK endpoint. Here, the number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*μg/mL
Arm/Group | SHP643 Prefilled Syringe (PFS) | SHP643 Autoinjector (AI)
Number analyzed (Participants) | 89 | 89
day*μg/mL | 352.5 (32.9) | 380.3 (40.8)
Statistical Analysis 1: Comparison: SHP643 Prefilled Syringe (PFS) vs SHP643 Autoinjector (AI); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio of Geometric least squares Means = 1.079, 90% CI 2-sided [0.987 to 1.179]

3. Primary Outcome: Maximum Observed Plasma Drug Concentration (Cmax) of SHP643 in Plasma
Description: Cmax is the maximum observed plasma concentration of SHP643 in Plasma was reported. Geometric mean and geometric coefficient of variation percent (CV%) was reported.
Time Frame: Pre-dose, 8, 24, 48, 72, 96, 168, 336, 504, 672, 1008, 1344, 2016, 2664 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (ug/mL)
Arm/Group | SHP643 Prefilled Syringe (PFS) | SHP643 Autoinjector (AI)
Number analyzed (Participants) | 94 | 94
microgram per milliliter (ug/mL) | 15.86 (40.6) | 18.35 (48.0)
Statistical Analysis 1: Comparison: SHP643 Prefilled Syringe (PFS) vs SHP643 Autoinjector (AI); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio of Geometric least squares Means = 1.157, 90% CI 2-sided [1.044 to 1.281]

4. Primary Outcome: Minimum Time to Reach (Tmax) in Maximum Observed Plasma Drug Concentration of SHP643 in Plasma
Description: Tmax of of SHP643 in plasma was reported.
Time Frame: Pre-dose, 8, 24, 48, 72, 96, 168, 336, 504, 672, 1008, 1344, 2016, 2664 hours post-dose
Population: PPK set was defined as all randomized participants who received the complete dose of SHP643 and had sufficient data to calculate at least one primary PK endpoint. Here, the number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: day
Arm/Group | SHP643 Prefilled Syringe (PFS) | SHP643 Autoinjector (AI)
Number analyzed (Participants) | 94 | 94
day | 4.00 [3.00 to 19.97] | 4.00 [2.00 to 6.92]

5. Primary Outcome: Terminal Half-Life (T1/2) of SHP643 in Plasma
Description: t1/2 of of SHP643 in plasma was reported.
Time Frame: Pre-dose, 8, 24, 48, 72, 96, 168, 336, 504, 672, 1008, 1344, 2016, 2664 hours post-dose
Population: as for outcome 2
Measure: Median (Full Range); unit: day
Arm/Group | SHP643 Prefilled Syringe (PFS) | SHP643 Autoinjector (AI)
Number analyzed (Participants) | 89 | 89
day | 13.76 [9.70 to 20.5] | 13.20 [8.21 to 40.1]

6. Primary Outcome: Apparent Total Body Clearance for Extravascular Administration Divided by the Fraction of Dose Absorbed (CL/F) of SHP643 in Plasma
Description: CL/F of of SHP643 in plasma was reported. Geometric mean and geometric coefficient of variation percent (CV%) was reported.
Time Frame: Pre-dose, 8, 24, 48, 72, 96, 168, 336, 504, 672, 1008, 1344, 2016, 2664 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per day (L/day)
Arm/Group | SHP643 Prefilled Syringe (PFS) | SHP643 Autoinjector (AI)
Number analyzed (Participants) | 89 | 89
liter per day (L/day) | 0.8511 (32.9) | 0.7888 (40.8)

7. Primary Outcome: Apparent Volume of Distribution Associated With the Terminal Slope Following Extravascular Administration Divided by the Fraction of Dose Absorbed (Vdz/F) of SHP643 in Plasma
Description: Vdz/F of SHP643 in plasma was reported. Geometric mean and geometric coefficient of variation percent (CV%) was reported.
Time Frame: Pre-dose, 8, 24, 48, 72, 96, 168, 336, 504, 672, 1008, 1344, 2016, 2664 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters (L)
Arm/Group | SHP643 Prefilled Syringe (PFS) | SHP643 Autoinjector (AI)
Number analyzed (Participants) | 89 | 89
Liters (L) | 16.79 (31.6) | 15.37 (42.7)

8. Primary Outcome: Terminal Elimination Rate Constant (Lambda z) of SHP643 in Plasma
Description: Lambda z of SHP643 in Plasma was reported. Geometric mean and geometric coefficient of variation percent (CV%) was reported.
Time Frame: Pre-dose, 8, 24, 48, 72, 96, 168, 336, 504, 672, 1008, 1344, 2016, 2664 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: one per day (1/day)
Arm/Group | SHP643 Prefilled Syringe (PFS) | SHP643 Autoinjector (AI)
Number analyzed (Participants) | 89 | 89
one per day (1/day) | 0.05070 (15.1) | 0.05132 (22.1)

9. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product that did not necessarily have a causal relationship with the investigational product (IP) or medicinal product. A treatment-emergent AE (TEAE) was defined as any event emerging or manifesting at or after the initiation of treatment with an IP or medicinal product or any existing event that worsened in either intensity or frequency following exposure to the IP or medicinal product.
Time Frame: From start of study drug administration up to Day 112 (End of Study/Early Termination [EOS/ET])
Population: Safety analysis set consisted of all randomized participants who received the dose of SHP643.
Measure: Count of Participants; unit: Participants
Arm/Group | SHP643 Prefilled Syringe (PFS) | SHP643 Autoinjector (AI)
Number analyzed (Participants) | 94 | 96
Participants | 19 | 30

10. Secondary Outcome: Number of Participants Who Developed Positive Antidrug Antibodies to SHP643 at Specified Time Points
Description: Plasma samples were analyzed for presence of antidrug antibodies to SHP643. Participants who developed positive results for SHP643 antibodies were reported.
Time Frame: Day 1, 14, 28, 56 and 112 (End of Study/Early Termination [EOS/ET])
Population: Safety analysis set consisted of all randomized participants who received the dose of SHP643.
Measure: Count of Participants; unit: Participants
Arm/Group | SHP643 Prefilled Syringe (PFS) | SHP643 Autoinjector (AI)
Number analyzed (Participants) | 94 | 96
Participants
  Participants with positive ADA: Day 1 | 1 | 0
  Participants with positive ADA: Day 14 | 0 | 0
  Participants with positive ADA: Day 28 | 1 | 0
  Participants with positive ADA: Day 56 | 0 | 1
  Participants with positive ADA: Day 112 (EOS/ET) | 0 | 1

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to Day 112 (End of Study/Early Termination [EOS/ET])
Arm/Group | SHP643 Prefilled Syringe (PFS) | SHP643 Autoinjector (AI)
All-Cause Mortality (participants affected / at risk) | 0/94 | 0/96
Serious Adverse Events (participants affected / at risk) | 2/94 | 2/96
Other Adverse Events (participants affected / at risk) | 0/94 | 9/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SHP643 Prefilled Syringe (PFS) (N=94) | SHP643 Autoinjector (AI) (N=96)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Abortion induced (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SHP643 Prefilled Syringe (PFS) (N=94) | SHP643 Autoinjector (AI) (N=96)
Injection site haemorrhage (General disorders) | 0 (0) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2019-01-29): https://cdn.clinicaltrials.gov/large-docs/39/NCT03918239/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-19): https://cdn.clinicaltrials.gov/large-docs/39/NCT03918239/SAP_001.pdf